CLINICAL TRIAL: NCT02324491
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial of ZGN-440 (Subcutaneous Beloranib in Suspension) in Obese Subjects With Type 2 Diabetes Mellitus to Evaluate Weight Reduction, Glycemic Control, Safety, and Tolerability
Brief Title: An Efficacy and Safety Study of Beloranib in Obese Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to analyze available safety and efficacy data
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZAF-203
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — CKD732

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ZGN-440 Injectable Suspension (1.2mg) (Experimental): ZGN-440 for Injectable Suspension
  Interventions: Drug: ZGN-440 for Injectable Suspension
- ZGN-440 Injectable Suspension (1.8mg) (Experimental): ZGN-440 for Injectable Suspension
  Interventions: Drug: ZGN-440 for Injectable Suspension
- Placebo (Placebo Comparator): ZGN-440 Placebo for Injectable Suspension
  Interventions: Drug: ZGN-440 Placebo for Injectable Suspension

INTERVENTIONS:
Drug: ZGN-440 for Injectable Suspension — Subjects will receive ZGN-440 twice weekly subcutaneous injections for up to 52 weeks.
  Other Names: Beloranib; ZGN-440
  Arms: ZGN-440 Injectable Suspension (1.2mg); ZGN-440 Injectable Suspension (1.8mg)
Drug: ZGN-440 Placebo for Injectable Suspension — Subjects will receive placebo twice weekly subcutaneous injections for up to 52 weeks.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of ZGN-440 (beloranib) in obese adult subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Phase 2, randomized, double-blind, placebo-controlled, parallel dose arms study with 12-month randomized treatment.

ELIGIBILITY:
Inclusion Criteria:

* Obese with BMI ≥30 kg/m2
* Type 2 diabetes mellitus
* HbA1c of 7-11%
* Fasting glucose <15.5 mmol/L
* Treated with diet and exercise alone or with a stable regimen of metformin, sulfonylurea, pioglitazone, DPP-4 inhibitor, GLP-1 receptor agonist, SGLT-2 inhibitor or any combination of these agents
* Female subjects must be surgically sterile, post-menopausal or using long-acting contraception, which includes intrauterine devices or use of an implanted or injectable contraceptive

Exclusion Criteria:

* Current or recent use of insulin
* Severe hypoglycemia within the prior 6 months
* Metabolic disorders or genetic disorders linked to obesity (e.g., Prader-Willi Syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to Week 26
Safety and tolerability assessed by adverse events, laboratory evaluations, ECGs, vital signs, physical examinations | Baseline to Week 26 and Week 52

SECONDARY OUTCOMES:
Change in body weight | Baseline to Week 52
Change in fasting glycemic parameters | Baseline to Week 26 and Week 52
  HbA1c, plasma glucose
Change in cardiometabolic parameters | Baseline to Week 26 and Week 52
  Blood pressure, lipid concentrations, hs-CRP
Change in Patient Reported Outcomes (PRO) scores | Baseline to Week 26 and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD, Study Director — Zafgen, Inc.
Locations (16):
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Pendlebury Research, Cardiff, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Illawara Diabetes Service, Wollongong, New South Wales
  - Q-Pharm, Herston, Queensland
  - Ipswich Research Institute, Ipswich, Queensland
  - AusTrials, Sherwood, Queensland
  - CMAX, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - Austin Health, Heidelberg West, Victoria
  - Emeritus Research, Malvern East, Victoria
  - Baker IDI Heart and Diabetes Institute, Melbourne, Victoria
  - Keogh Institute for Medical Research, Nedlands, Western Australia

REFERENCES:
- [Derived] Proietto J, Malloy J, Zhuang D, Arya M, Cohen ND, de Looze FJ, Gilfillan C, Griffin P, Hall S, Nathow T, Oldfield GS, O'Neal DN, Roberts A, Stuckey BGA, Yue D, Taylor K, Kim D. Efficacy and safety of methionine aminopeptidase 2 inhibition in type 2 diabetes: a randomised, placebo-controlled clinical trial. Diabetologia. 2018 Sep;61(9):1918-1922. doi: 10.1007/s00125-018-4677-0. Epub 2018 Jul 11. PMID 29992370